CLINICAL TRIAL: NCT04741399
Title: EXperienceS and aTtitudes Towards Agitated Behaviours in Tbi ICu Patients (EXSTATIC): a Protocol for an Interprofessional Mixed-method Study
Brief Title: Experiences and Attitudes Towards Agitated Behaviours in TBI ICU Patients: a Protocol for an Interprofessional Mixed-method Study
Acronym: EXSTATIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Centre Universitaire de Santé McGill (Unknown)
Responsible Party: Sponsor
Other Study IDs: MP-32-2021-2198
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Trauma Injury; Intensive Care Neurological Disorder
Keywords: Agitation; Healthcare professionals
MeSH Terms: conditions — Accidental Injuries; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EXSTATIC is a multicenter mixed methods convergent study exploring experiences and attitudes of ICU healthcare professionals caring of agitated traumatic brain injury (TBI) patients. The study aims to explore the experiences and attitudes of ICU nurses and other ICU healthcare professionals on the management of agitation in acute TBI patients. This project includes three qualitative methods and one quantitative method. First step consists in structured observations of the daily routine of ICU healthcare professionals when TBI patient admitted in the ICU develops agitation. This step will allow us to raise emerging research questions from the field and to develop subsequent steps. Secondly, we will conduct semi-structured interviews with ICU nurses. Themes emerged in the interviews are essential to understand nurses' experiences and attitudes towards TBI agitated patients and describe their relational role amongst patients, other professionals and families. A retrospective cohort of TBI patients gathered through medical files will follow aiming to document in which way observations in the two first phases are reflected in the clinical notes. Finally, different ICU healthcare professionals will be invited to participate in focus groups to identify further themes in semi-structured interviews in nurses, compare them and prioritize which are the most relevant to nurses experiences and which ones need to be addressed for their future practice. The integration of the different methods will be done using sequential steps of the research (the previous informing the next one) and by the integration of results for each step. Qualitative data will be evaluated following the grounded theory using thematic analysis. Quantitative data will be analysed using descriptive statistics. Qualitative and quantitative results will be combined in a convergent interactive interpretative design. Race and gender perspective will be integrated in collection, analysis and interpretation of data.

DETAILED DESCRIPTION:
A convergent design will be performed using three qualitative research methods (structured observations, semi-structured interviews and focus groups) and a quantitative research method (retrospective observational study).

First, a researcher will observe the daily ICU routine, in two ICU units, when a TBI-patient is admitted. In this first step, the specific objective is to observe the care of TBI patients during periods of agitation, to understand how it affects the actions of healthcare professionals and their interactions with each other and other actors present in the unit. These observations will enable researchers to detect non-verbal expression of feelings, interactions and communication between patients, their family and health professionals as well as interactions between health professionals at the bedside. The observations will also enable us to map bedside clinical activities made by health professionals and the time spent doing them. The goal is to develop a repertoire of situations combining the degree of agitation, the resources present, the experience and the effects on the staff, the patient and their relatives, the actions and medical decisions in response to agitation. The data gathered in this phase will inform the interview guide for the semi-structured interviews.

In the second phase, we will conduct semi-structured interviews with ICU nurses to explore their experiences and attitudes towards the care of TBI patients with agitated behaviours. Nurses will be interviewed as they are the healthcare professionals most present at the bedside of TBI patients and their families. Semi-structured interviews enable to explore nurse's perspectives and experiences. This will also allow us to investigate how these experiences can predict their reactions to agitated behaviours, and how these reactions are shared between different health professionals or also with hospital health personnel. This particular phase enables us to uncover unanticipated themes.

We will then undertake a retrospective observational study aiming to describe the documentation of agitated behaviours in TBI patients and interventions to manage them. In this step, the objective is to substantiate the documentation of the significant elements identified in the first two phases of the study. This third phase will be complementary to the previous two phases and will allow to document in which way observations in the first two phases are reflected in the clinical notes. A convenience sample of consecutive admissions for TBI with an abnormal CT-scan will be reviewed.

Finally, interprofessional focus groups will be conducted in order to gain insights into ICU healthcare professionals experiences and explore their attitudes and needs when TBI patients develop agitation. Group process can help people to explore and clarify their views and to share ideas and perceptions. All healthcare professional who participate in the care of TBI patients in the ICU will be solicited for participation. Specifically, the aim is to discuss the various themes identified in the previous steps and understand their relational dimension among different healthcare professionals.

The integration of the different methods will be done by the connection of the different steps and by the integration of results for each step. This multistep approach allows to identify organizational, cultural factors and to better understand social interactions as well as health care delivery process.

ELIGIBILITY:
Inclusion Criteria:

* All professionals belonging to the intensive care team (nurses, occupational therapists, beneficiary attendants, ICU physicians, physiotherapists, respiratory therapists, pharmacists, unit coordinators), employed full-time or part-time in any shift with a minimum of 1 year of trauma intensive care experience can be included to participate in the semi-structured interviews and focus groups
* All patients suffering from a TBI with an abnormal CT scan admitted to the ICU will be included for the structured observation
* In the retrospective observational study, a convenience sample of 25 patients per centre (50 patients in total) admitted six months before the observational period will be included for data collection.

Exclusion Criteria:

* Temporary staff, students or residents will be excluded from semi-structured interviews and focus groups

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: ICU healthcare professionals ICU TBI patients
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
To explore the experiences and attitudes of the healthcare professionals managing agitation of TBI patients in two ICUs of level-1 Canadian trauma hospitals | December 2020-October 2021
  To unveil the perceptions, the practices, the consequences and the risks of handling TBI agitated patients.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saavedra-Mitjans M, David PM, Frenette AJ, Arbour C, Perreault M, Williams V, Bernard F, Williamson D. EXperienceS and aTtitudes towards Agitated behaviours in Traumatic brain injury in the Intensive Care unit patients (EXSTATIC): a protocol for an interprofessional mixed-method study. BMJ Open. 2021 Jul 14;11(7):e045816. doi: 10.1136/bmjopen-2020-045816. PMID 34261680